CLINICAL TRIAL: NCT04060381
Title: Myocardial Deformation Before and After Birth, and Under Altered Preload, Afterload and Heart Rate in New-borns
Brief Title: Myocardial Deformation Before and After Birth
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Gottfried Greve, Consultant/ Professor, Haukeland University Hospital
Other Study IDs: 2015/1918
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Dysfunction; Newborn Morbidity; Maternal Obesity
Keywords: Spackle tracking echocardiography; Tissue doppler; Neonates; Infants; Maternal obesity
MeSH Terms: conditions — Pregnancy in Obesity | interventions — Blood Transfusion; Ibuprofen; Epinephrine; Norepinephrine; Dopamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Fetuses of normal weight women: Fetuses of normal pregnancies of normal weight mothers are included from gestational week 37
- Fetuses of severely obese women: Fetuses of normal pregnancies of severly obese mothers are included from gestational week 37
- New-borns in need of blood transfusion: Neonates mainly receive blood due to blood loss, often because of repeated blood sampling
  Interventions: Drug: Blood transfusion, Ibuprofen, or epinephrine, norepinephrine or dopamine
- New-borns in need for closure of the arterial duct: Neonates mainly receive medication (Ibuprofen) because of symptoms like apnea, due to their patent arterial duct.
  Interventions: Drug: Blood transfusion, Ibuprofen, or epinephrine, norepinephrine or dopamine

INTERVENTIONS:
Drug: Blood transfusion, Ibuprofen, or epinephrine, norepinephrine or dopamine — Treatment/ intervention given according to standard protocols at the Neonatal Intensive Care Unit
  Other Names: Volume treatment; Blood pressure elevation
  Groups: New-borns in need for closure of the arterial duct; New-borns in need of blood transfusion

SUMMARY:
Knowledge on the changes in myocardial function in the last weeks before birth and during the first year of life is limited. Through fetal and post-natal echocardiography we intend to describe these changes using myocardial tissue recognition techniques (Speckle tracking echocardiography and Tissue Doppler echocardiography) in healthy neonates, born to term of healthy women after uncomplicated pregnancies. We will compare the findings in this cohort to a cohort of neonates born to term of women with severe pre-pregnancy obesity.

Sick neonates in intensive care units with various cardiac and non-cardiac conditions are often exposed to treatment that may affect both their cardiac function and important echo-variables per se. Using echocardiography, we will examine these changes in neonates treated with blood transfusion, catecholamines and in those treated with Ibuprofen due to a haemodynamic significant arterial duct.

DETAILED DESCRIPTION:
Before, during and after birth major changes take place in the cardiovascular system. The last weeks prior to birth there is an oxidative stress and after birth, there is normally a large step up in blood oxygen tension when the lungs take over oxidation of the blood. Simultaneously there are changes in the vascular resistance in both the pulmonary- and systemic part of the circulation and ductus venous, the arterial duct, and foramen ovale close. Combined these will significantly alter the physical conditions under which the myocardium is supposed to work.

This project will have five arms, all based on measurements of myocardial function and coronary perfusion by speckle tracking echocardiography (STE) in the last trimester of the pregnancy and in newborns with different gestational age and in sick newborns where myocardial function is affected by medical treatment or is an important part of the clinical situation.

1. Obtaining normal values for strain during the last trimester of the pregnancy and the first days after birth in child born to term.

   Hypothesis: After birth, there will be higher STE values in the left ventricle than before birth. This will increase further the first days post-partum in parallel with an altered hemodynamic situation and oxygen demand of the infant. The STE changes will take place at the same time, as there is an increased Doppler velocity in the aorta, the pulmonary artery and the coronary arteries

   Mothers (N= 150) will be recruited when they are coming to a routine fetal ultrasound scan. It will be made an echo-examination once per week from week 37 until birth. After birth the degree of placental transfusion (late cord clamping or not) will be noticed. Ventricular size, Doppler velocities in the ascending aorta and pulmonary artery, STE and coronary flow during the first three days of life and one year of age will be assessed
2. Evaluate the effect of maternal obesity on cardiac function in newborns up to one year of age.

   Hypothesis: Maternal sever obesity will result in reduced cardiac function in their neonates. However, cardiac function will normalize within the first year of life. A reduction in afterload will reduce strain measured by STE and coronary.

   Mothers (N=75) with sever obesity will be recruited from the outpatient clinic for obese women. First day after birth, the newborn will have a comprehensive echocardiographic examination within the first few hours, then the two following days, at the day equivalent to gestational age 42+0 weeks and finally at 1 year of age. Cardiac morphology, ventricular sizes and Doppler velocities in the ascending aorta and pulmonary artery as well as a strain measured by STE for both ventricles will be assessed. Fetal malformations or diseases will result in exclusion from the study.
3. Measuring deformation when preload is increased by intravenous fluid treatment and blood transfusion Hypothesis: Increased preload in the form of saline infusion or blood transfusion will result in a temporary increase of STE and coronary blood flow.

   Newborns (N=25 blood transfusion and 25 NaCl-infusion) who need infusion of sodium chloride (NaCl 9mg) / ml or transfusion of packed red blood cellssuspended in 100 mL of saline- adenine-glucose-mannitol (SAGMAN) will be recruited. To obtain rehydration or optimization of intravascular volume it is common to provide NaCl 9 mg/ml, 10-20 ml/kg in 10-120 minutes. Blood transfusion is used in severe anemia and hemolytic diseases. The regular blood transfusion dose is SAGMAN packed red blood cells10-15ml/ kg body weight over 2-3 hours. Children requiring exchange transfusion, with heart failure or congenital heart defects will be excluded.
4. Measuring deformation when afterload and heart rate are increased during infusion of catecholamines.

   Hypothesis: Dopamine, epinephrine and/ or nor-epinephrine will increase heart rate and blood pressure and due to this increase the strain measured by STE, coronary blood flow, and Doppler velocity in the aorta pulmonary artery.

   Newborns (N=25) who need dopamine (2.5 to 15 ug/kg /min iv.) and or epinephrine / nor-epinephrine to maintain an adequate blood pressure will be recruited. Only children where an echo-exam before starting treatment is possible will be recruited. If the treatment does not achieve a rise in the blood pressure above the 2.5 percentile for gestational age, the baby will be excluded.
5. Measuring deformation when afterload (volume) is reduced following pharmacological closure of a patent ductus arteriosus.

Hypothesis: A reduction in afterload will reduce strain measured by STE and coronary.

Patients (N=25) with a suspected patent ductus arteriosus (PDA) are always referred to echocardiography before starting treatment with Indomethacin and after the treatment has stopped. Present clinical procedures for closure of the ductus will be followed, . Time of echocardiography will be standardized to just before and at least 12 hours after the last dose of Ibuprofen has been provided (t½ ≈ 2.5-11 hrs.).

ELIGIBILITY:
Inclusion Criteria:

* Normal pregnancies
* Newborns in need of blood transfusion
* Newborns in need of medical closure of the arterial duct
* Maternal obesity

Exclusion Criteria:

* Abnormal pregnancies except maternal obesity
* Congenital heart defects
* Other malformation syndromes

Max Age: 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Either recruited during pregnancies or as newborns
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in myocardial function | Maximum 1 year and 5 weeks
  Per cent change in longitudinal global strain

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Eventually strain data.